CLINICAL TRIAL: NCT04524507
Title: IGHID 12021 - A Randomized, Phase II Study Comparing the Efficacy and Safety of Standard Versus High-Titer Anti-Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Neutralizing Antibody Plasma in Hospitalized Patients With COVID-19
Brief Title: Coronavirus Disease 2019 (COVID-19) Antibody Plasma Research Study in Hospitalized Patients
Acronym: UNC CCP RCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20-1544
Record Dates: First submitted 2020-08-21; First posted 2020-08-24 (Actual); Results first posted 2021-11-23 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-06

CONDITIONS: COVID-19
Keywords: COVID-19; Coronavirus; Infection; SARS-CoV-2; Randomized; Hospitalized; Plasma; Neutralizing; Antibody
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Infections | interventions — tyrosyltubulin carboxypeptidase

STUDY DESIGN:
Intervention Model Description: This study has 2 treatment arms and participants will be assigned/randomized to one arm:
  1. CCP1 - CCP tested for the presence of anti-SARS-CoV-2 antibodies and assigned high-titer
  2. CCP2 - CCP tested for the presence of anti-SARS-CoV-2 antibodies and assigned standard-titer
Who Masked: Participant, Investigator
Masking Description: This study is double-blinded so neither the participant nor the study team/investigators will know which plasma treatment (CCP1 or CCP2) that the participant is receiving.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- High-Titer (CCP1) (Experimental): Within 8 days of COVID symptom onset and no more than 48 hours following hospitalization, participants will be randomized to and receive high-titer ABO-compatible convalescent COVID-19 plasma (CCP1) within 24 hours following random assignment.
  Interventions: Biological: High-titer Convalescent COVID-19 Plasma (CCP1)
- Standard-Titer (CCP2) (Active Comparator): Within 8 days of COVID symptom onset and no more than 48 hours following hospitalization, participants will be randomized to and receive standard-titer ABO-compatible convalescent COVID-19 plasma (CCP2) within 24 hours following random assignment.
  Interventions: Biological: Standard-titer Convalescent COVID-19 plasma (CCP2)

INTERVENTIONS:
Biological: High-titer Convalescent COVID-19 Plasma (CCP1) — At least two units of CCP transfused 4-24 hours apart on Study Day 0. A third unit may be administered, if available.
  Arms: High-Titer (CCP1)
Biological: Standard-titer Convalescent COVID-19 plasma (CCP2) — At least two units of CCP transfused 4-24 hours apart on Study Day 0. A third unit may be administered, if available.
  Arms: Standard-Titer (CCP2)

SUMMARY:
The purpose of this research study is to find out if CCP is safe and to determine the safest and most effective level of anti-viral antibody when given to people admitted to the hospital with confirmed COVID-19 infection. Participants enrolled on this study will be transfused with 2 units of CCP through an IV. These units will be given one at a time 4 to 24 hours apart. Participants will be randomized to receive either 2 units with standard antibody levels as recommended by the FDA or 2 units with an antibody level higher than that recommended by the FDA. This study is experimental and CCP is investigational and has not been approved by the FDA for the treatment of COVID-19. The CCP is collected per FDA guidelines from persons recovered from COVID-19 infection. The plasma contains antibodies and possibly other properties that inhibit the virus. The investigators do not know if the level of antibodies present in the CCP will make a difference in how the participant's body is able to fight the infection and hope to learn that in this study.

DETAILED DESCRIPTION:
This randomized, double-blinded, phase 2 trial will assess the efficacy and safety of anti-SARS-CoV-2 convalescent plasma in hospitalized patients with less than 8 days of symptoms. Eligible participants will receive institutional-guided standard-of-care (SOC) and ABO-compatible convalescent COVID-19 plasma (CCP). The CCP units will be tested for the presence of anti-SARS-CoV-2 antibodies and pre-assigned as high-titer (CCP1) or standard-titer (CCP2) in a 1:1 randomization. Participants and clinical investigators will be blinded to the CCP titer group identities.

The investigators plan to enroll approximately 56 participants (28 in each group) at UNC-Chapel Hill. Participants will be randomized within 48 hours of admission to a COVID service and will receive convalescent plasma within 24 hours of randomization. At least two units of CCP will be transfused 4-24 hours apart on study Day 0. If available, a third unit may be administered. All participants will undergo a series of safety and efficacy assessments pre-, during, and post-transfusion. Samples for research will be collected on Day 0 through Day 28, unless previously discharged. Additionally, after discharge, participants can provide longitudinal samples collected at 1, 3, and 6-month timepoints after the infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Age at least 18 years
2. Ability and willingness of participant or Legally Authorized Representative (LAR) to give written informed consent.
3. Laboratory confirmed diagnosis of infection with SARS-CoV-2 by PCR
4. Hospitalized for COVID-19 with one or more respiratory or gastrointestinal (GI) symptoms:

   * COVID-19 associated respiratory symptoms include but are not limited to: cough, shortness of breath, difficulty breathing, or sore throat
   * COVID-19 associated GI symptoms include but are not limited to: loss of taste, loss of sense of smell, diarrhea, nausea, or vomiting,

Note: Respiratory and GI symptoms other than those listed above, must be noted as acceptable and signed by study PI or designee.

Exclusion Criteria:

1. Receipt of pooled immunoglobulin in past 30 days
2. Current or prior enrollment in a SARS-CoV-2 antibody or T-cell therapeutic study.

   Note: Patients enrolled on other randomized controlled trials of pharmaceutical and/or non-pharmaceutical interventions for COVID and meeting eligibility criteria will not be excluded, as determined by study PI (or designee) on a case-by-case basis and as allowed by eligibility criteria of the other trials.
3. Contraindication to transfusion or history of prior reactions to transfusion blood products. This may include religious or cultural objections to receiving blood products and transfusions.
4. ABO-compatible titered plasma is not available
5. > 10 days from noted COVID-related subjective or objective fever at randomization. Patients without subjective or objective fever, > 10 days from symptom onset as determined by study PI.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2020-08-27 (Actual); Primary Completion 2021-01-04 (Actual); Study Completion 2021-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luther A Bartelt, MD, Principal Investigator — UNC-Chapel Hill; David M Margolis, MD, Principal Investigator — UNC-Chapel Hill
Locations (1):
- University of North Carolina Health Care, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual data that supports the results will be shared beginning 12 to 24 months following publication provided the investigator/researcher who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, Analytic Code
Time Frame: 12-24 months after publication
Access Criteria: Investigators/researchers who propose to use study data will need to have IRB, IEC, or REB approval and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Derived] Bartelt LA, Markmann AJ, Nelson B, Keys J, Root H, Henderson HI, Kuruc J, Baker C, Bhowmik DR, Hou YJ, Premkumar L, Cornaby C, Schmitz JL, Weiss S, Park Y, Baric R, de Silva AM, Lachiewicz A, Napravnik S, van Duin D, Margolis DM. Outcomes of Convalescent Plasma with Defined High versus Lower Neutralizing Antibody Titers against SARS-CoV-2 among Hospitalized Patients: CoronaVirus Inactivating Plasma (CoVIP) Study. mBio. 2022 Oct 26;13(5):e0175122. doi: 10.1128/mbio.01751-22. Epub 2022 Sep 22. PMID 36135380

RESULTS

PARTICIPANT FLOW:
Groups:
- High-Titer (CCP1): Within 10 days of COVID symptom onset and no more than 48 hours following hospitalization, participants will be randomized to and receive high-titer ABO-compatible convalescent COVID-19 plasma (CCP1) within 24 hours following random assignment.
  High-titer Convalescent COVID-19 Plasma (CCP1): At least two units of CCP transfused 4-24 hours apart on Study Day 0. A third unit may be administered, if available.
- Standard-Titer (CCP2): Within 10 days of COVID symptom onset and no more than 48 hours following hospitalization, participants will be randomized to and receive standard-titer ABO-compatible convalescent COVID-19 plasma (CCP2) within 24 hours following random assignment.
  Standard-titer Convalescent COVID-19 plasma (CCP2): At least two units of CCP transfused 4-24 hours apart on Study Day 0. A third unit may be administered, if available.
Period: Overall Study
Arm/Group | High-Titer (CCP1) | Standard-Titer (CCP2)
Started | 15 | 41
Received Intervention | 14 | 41
Hospital Discharge (Discharged at or before Day 28.) | 13 | 27
Completed (Day 28) | 9 | 18
Not Completed | 6 | 23
Not completed — Lost to Follow-up | 2 | 4
Not completed — Withdrawal by Subject | 2 | 9
Not completed — Death | 2 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High-Titer (CCP1) | Standard-Titer (CCP2) | Total
Number analyzed (Participants) | 15 | 41 | 56
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 57 [49 to 75] | 62 [54 to 67] | 61 [52.5 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 14 | 20
  Male | 9 | 27 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 13 | 18
  Not Hispanic or Latino | 10 | 27 | 37
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 12 | 14
  White | 8 | 15 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 13 | 18
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 41 | 56

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Serious Adverse Events (SAE) Through Study Day 14
Description: Total number of SAE among all participants through Day 14; Definition of SAE per protocol and will only be included if related to COVID-19 Convalescent Plasma (CCP): 1. Death; 2. Life-threatening (immediate risk of death); 3. Prolongation of existing hospitalization; 4. Persistent or significant disability or incapacity; OR 5. Important medical events that may not result in death, be life threatening, or require intervention or escalation of care may be considered a serious adverse event when, based upon appropriate medical judgment, they may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias, or convulsions that do not result in inpatient hospitalization.
Time Frame: 14 days
Measure: Number; unit: Serious Adverse Events
Arm/Group | High-Titer (CCP1) | Standard-Titer (CCP2)
Number analyzed (Participants) | 14 | 41
Serious Adverse Events | 0 | 0

2. Primary Outcome: Median Time to Hospital Discharge (or Discharge Equivalent) Following First Dose of CCP
Description: Median number of days to hospital discharge following first dose of CCP among all participants.
Time Frame: up to 28 days
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | High-Titer (CCP1) | Standard-Titer (CCP2)
Number analyzed (Participants) | 14 | 41
Days | 5 [2 to 6] | 7 [3 to 20]

ADVERSE EVENTS:
Time Frame: From the time participants received the study intervention through Day 28.
Arm/Group | High-Titer (CCP1) | Standard-Titer (CCP2)
All-Cause Mortality (participants affected / at risk) | 2/14 | 10/41
Serious Adverse Events (participants affected / at risk) | 2/14 | 15/41
Other Adverse Events (participants affected / at risk) | 13/14 | 38/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High-Titer (CCP1) (N=14) | Standard-Titer (CCP2) (N=41)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 10 (13)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 2 (2)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Acute respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High-Titer (CCP1) (N=14) | Standard-Titer (CCP2) (N=41)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 4 (7)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 7 (8) | 14 (18)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 14 (18)
Aspartate aminotransferase increased (Investigations) | 4 (5) | 7 (8)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 4 (4)
Bacteremia (Infections and infestations) | 0 (0) | 3 (3)
Blood albumin decreased (Investigations) | 1 (1) | 5 (5)
Blood bicarbonate decreased (Investigations) | 0 (0) | 3 (3)
Blood bilirubin increased (Investigations) | 0 (0) | 6 (8)
Blood creatinine increased (Investigations) | 2 (2) | 4 (4)
Blood potassium decreased (Investigations) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 4 (5)
Bradycardia (Cardiac disorders) | 1 (1) | 2 (2)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 2 (2) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 7 (7)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (2) | 10 (11)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 7 (7)
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 7 (11)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (4) | 11 (13)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Hyponatremia (Metabolism and nutrition disorders) | 4 (4) | 9 (9)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
International normalized ratio increased (Investigations) | 0 (0) | 7 (9)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Lymphocyte count decreased (Investigations) | 2 (2) | 11 (13)
Neutrophil count decreased (Investigations) | 1 (1) | 2 (2)
Platelet count decreased (Investigations) | 1 (1) | 1 (3)
Pneumonia (Infections and infestations) | 1 (1) | 4 (5)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 3 (4)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
White blood cell count decreased (Investigations) | 0 (0) | 3 (3)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Venous occlusion (Vascular disorders) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 4 (4)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-18): https://cdn.clinicaltrials.gov/large-docs/07/NCT04524507/Prot_SAP_000.pdf